CLINICAL TRIAL: NCT00927108
Title: Adult Neuronal Progenitor Stem Cell Project
Brief Title: Rajavtihi Neuronal Adult Stem Cells Project
Acronym: RNASc
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Collaborators: Rajavithi Biomolecular Research Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RH-CMR-005
Record Dates: First submitted 2009-06-22; First posted 2009-06-24 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Alzheimer's Disease; Parkinson's Disease; Multiple Sclerosis
Keywords: Adult Progenitor Stem cells; Alzheimer's disease; Parkinson's disease; Multiple sclerosis
MeSH Terms: conditions — Alzheimer Disease; Parkinson Disease; Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Cell culture
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Progenitor Stem Cell Culture

SUMMARY:
To study the success of Oligodendrocyte progenitor cell culture project in Rajavithi Hospital to identify an unlimited clone human neuronal progenitor stem cells from the human brain in the Biomolecular Research Center. This study aims to produce the reproductive clone of neuronal development protocols and advance projects. Neuronal cells such as pyramidal cells, oligodendrocyte, and dopaminergic neuron differentiation protocol/projects for treatment of Alzheimer's disease, Multiple sclerosis, and Parkinson's disease respectively in next phase of clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have elective craniotomy or.
* Patients who have elective ventriculostomy surgery or.
* Patients who have elective muscle biopsy or nerve biopsy.
* Patient who have emergency craniectomy for life threatening from emergency medical and surgical conditions such as Brain herniation or head injury

Exclusion Criteria:

* Central nervous system infection for example tuberculous or any bacterial infection, Viral infection, fungal infection.
* Central nervous system Tumor, Malignancy and metastasis.

Ages: 20 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Subsai Kongsaengdao, M.D., Principal Investigator — Department of Medical Services Ministry of Public Health of Thailand
Locations (1):
- Rajavithi Hospital, Bangkok, Thailand